CLINICAL TRIAL: NCT01282671
Title: Effects of Deep Breathing Exercises Two Months After Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government); Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Elisabeth Westerdahl, PhD, RPT, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Multic-PEP 2007-160
Record Dates: First submitted 2010-12-06; First posted 2011-01-25 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: CABG; Valve Surgery
Keywords: breathing exercises; cardiac surgery; lung function; postoperative complication; positive expiratory pressure
MeSH Terms: conditions — Postoperative Complications | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breathing exercises (Experimental): On the fourth postoperative day the patients are randomly assigned to a Treatment group continuing to perform deep breathing exercises for 2 months postoperatively and to a Control group who will perform no breathing exercises after the third postoperative day. Patient management is otherwise similar in the groups. The patients in the Deep breathing group will be instructed to perform breathing exercises (3 x 10 deep breaths) 5 times a day (document compliance) during the two postoperative months.
  Interventions: Other: Breathing exercises
- Control group (No Intervention): No breathing exercises.

INTERVENTIONS:
Other: Breathing exercises — On the fourth postoperative day the patients are randomly assigned to a Treatment group continuing to perform deep breathing exercises for 2 months postoperatively and to a Control group who will perform no breathing exercises after the third postoperative day. Patient management is otherwise similar in the groups. The patients in the Deep breathing group will be instructed to perform breathing exercises (3 x 10 deep breaths) 5 times a day (document compliance) during the two postoperative months. A Positive expiratory pressure (PEP) device PEP ventil, System 22 (Rium Medical, Täby, Sweden) is used to create an expiratory resistance of +10 cm H2O.
  Other Names: Intervention group: Performing breathing exercises.; Control group: No breathing exercises.
  Arms: Breathing exercises

SUMMARY:
Hypothesis: Deep breathing exercises performed during the first two months after cardiac surgery, will improve pulmonary function and patient-perceived quality of recovery.

Specific aim: To evaluate the effectiveness of breathing exercises performed with a mechanical device for positive expiratory pressure during the first two months after cardiac surgery compared to a control group performing no breathing exercises.

Design: A prospective, randomized, controlled two-center study.

DETAILED DESCRIPTION:
Contribution: The study will be taken place at two University hospitals in Sweden.

Uppsala university hospital (PhD, Registered physical therapist (RPT)) Margareta Emtner and RPT Charlotte Urell) and Örebro university hospital; (Elisabeth Westerdahl and RPT Marcus Jonsson).

Time planning: Application to the Research Ethics Committee april 2007. Data collection 2007-2011. Statistical analysis and manuscript writing 2011.

ELIGIBILITY:
Inclusion Criteria:

* A sample of 360 adults (>18 years) patients undergoing cardiac surgery at the two University hospitals are invited to participate in the study.
* Type of cardiac surgery included will be Coronary artery bypass graft surgery (CABG) with saphenous vein grafts and/or internal mammary artery graft, valve surgery or combinations of CABG and valve surgery.

Exclusion Criteria:

* Patients who have an emergency operation, previous cardiac or lung surgery, renal dysfunction requiring dialysis or are unable to communicate in Swedish will not be included.
* Patients who requires more than 24 hours respirator treatment, reintubation, reoperation, sternum instability/infection or develop a neurological, mental or haemodynamic complication that affects the patients' ability to collaborate, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2007-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Lung function measured as Forced expiratory volume in 1 second (FEV1) | Two months after surgery
  Spirometry is performed preoperatively and 2 months after surgery at the Departments of Clinical Physiology. A Jaeger MasterScreen Pulmonary functiontest (PFT)/Bodybox will be used at the University hospitals in Uppsala and Örebro. The medical laboratory technologists are blinded to the patient's treatment allocation. Static and dynamic lung volumes will be measured.

SECONDARY OUTCOMES:
Postoperative quality of recovery | Two months postoperatively
  Physical activity, postoperative pain, day of discharge, signs of pneumonia or pulmonary comlications will be noted. Patient-perceived quality of recovery will be assessed using a translated version of a recently validated quality of recovery score (QoR-40) designed to measure the patient's health status after surgery and anaesthesia. The SF (short form) -36 (first version) will be used for assessment of quality of life aspects.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Westerdahl, PhD, RPT, Principal Investigator — Region Örebro County
Locations (2):
- Sweden (2):
  - Uppsala University, Uppsala
  - Örebro University Hospital, Örebro, Örebro County

REFERENCES:
- [Result] Westerdahl E, Urell C, Jonsson M, Bryngelsson IL, Hedenstrom H, Emtner M. Deep breathing exercises performed 2 months following cardiac surgery: a randomized controlled trial. J Cardiopulm Rehabil Prev. 2014 Jan-Feb;34(1):34-42. doi: 10.1097/HCR.0000000000000020. PMID 24280904
- [Result] Jonsson M, Urell C, Emtner M, Westerdahl E. Self-reported physical activity and lung function two months after cardiac surgery--a prospective cohort study. J Cardiothorac Surg. 2014 Mar 28;9:59. doi: 10.1186/1749-8090-9-59. PMID 24678691